CLINICAL TRIAL: NCT05273970
Title: Electrochemical and Electrophysiological Correlates of Human Cognition, Emotion, and Behavior
Brief Title: Electrochemical and Electrophysiological Study
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arizona (Other)
Collaborators: Arizona State University (Other); Virginia Polytechnic Institute and State University (Other)
Responsible Party: Principal Investigator, Robert Bina, Assistant Professor - Neurosurgery, University of Arizona
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY00000295
Record Dates: First submitted 2022-02-28; First posted 2022-03-10 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Cognition; Medically Intractable Epilepsy
Keywords: epilepsy monitoring; seizure localization; neurotransmitters; electrophysiological parameters; Electrochemical gradients; Fast Scan Cyclic Voltammetry; SEEG

STUDY DESIGN:
Intervention Model Description: Recordings will be obtained from intracranial electrodes placed for clinical or approved research purposes during neurosurgical procedures, and/or thereafter, while patients are followed in the epilepsy monitoring unit (EMU). Electrodes approved for human use may be placed on the cortex or within subcortical structures. Recordings may be obtained during passive conditions and task-based recordings designed to study particular regions of interest will be carried out in the EMU, as well as passive without task performance.
  Patients undergoing surgery for invasive functional brain mapping may also undergo electrical microstimulation in addition to neurophysiological recording. Stimulation is typically delivered in 2-5 second bursts (25-50 Hz, 0.3 ms pulse width, 1-15 mA). Recording and microstimulation may take place either intra-operatively and/or post-operatively in the EMU.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Behavioral testing under intracranial monitoring (Experimental): Patients will undergo behavioral tasks while being monitored by intercranial electrodes
  Interventions: Other: Behavioral testing under intracranial monitoring

INTERVENTIONS:
Other: Behavioral testing under intracranial monitoring — After standard of care surgery to implant the electrodes is complete and patients have have recovered satisfactorily from the procedure, they will be asked to perform some computer based tasks to answer questions about pretend financial decisions, pay attention to certain images, watch videos, look at images, listen to sounds, or move a joystick.

SUMMARY:
This study will utilize computerized algorithms in combination with real-time intracranial neurophysiological and neurochemical recordings and microstimulation to measure cognitive and affective behavior in humans.

Questionnaires or simple behavioral tasks (game-like tasks on a computer or an iPad) may also be given to additionally characterize subjects on related cognitive or affective components. Importantly, for the purposes of understanding the function of the human brain, neural activity can be recorded and probed (i.e. microstimulation) while subjects are performing the same computerized cognitive and affective tasks. These surgeries allow for the in vivo examination of human neurophysiology and are a rare opportunity for such research.

The questionnaires and assessments proposed will provide insights into disorders (and anxiety, depression) and psychological status that we hope to understand in relation to the neurochemistry measures. They will also provide baseline information that may be used to characterize and group the population to further refine our understanding of the neural responses.

In addition to computerized testing, we plan to characterize subjects' behavior on related cognitive or affective components. Some neuropsychological questionnaires, many of which are administered for clinical reasons, may also be given to patients and healthy control subjects.

All patients undergoing epilepsy surgery or deep brain stimulation undergo a standard clinical neuropsychological battery to assess aspects of cognitive function. This is a regular aspect of their clinical assessment carried out prior to consideration for study inclusion. All participants are selected uniformly because they are undergoing surgery for intracranial electrode implantation. No particular ethnic group or population is targeted by or excluded from the study.

Those to be considered for inclusion in the proposed study performing more than 2 standard deviations below the mean on any aspect of cognitive functioning as determined by standard preoperative neuropsychological testing will be excluded from the study.

DETAILED DESCRIPTION:
Dysfunction in neurotransmission and neurophysiology can result in a range of psychiatric conditions including depression, anxiety, chronic pain, addiction disorders, and problems with attention (attention deficit disorder) and arousal (narcolepsy). Despite the clear importance of these neuromodulatory systems, practically nothing is known about how these systems act in real time (at sub-second timescales) in the human brain. This temporal resolution has proven to be important in basic research in rodent model organisms, where it has been shown that the extracellular concentration of neurotransmitters and neural electrophysiology changes within 100s of milliseconds of interacting with relevant stimuli while navigating moment-to-moment changes in the environment. Measurements with this kind of precision are necessary to be able to investigate how rapid changes in each of these signals modulate brain function, cognition, learning, mood, and behavior in humans.

Clinical context of proposed research: Patients with treatment (medication) resistant epilepsy can become candidates for surgical ablation of the epileptic foci. To determine which region of the brain is the source of the seizures, patient undergo phase-I and, if necessary, phase-II epilepsy monitoring. Phase-I requires non-invasive electroencephalographic recordings using electrodes placed on the patient's scalp. If these recordings are inconclusive, a patient becomes a candidate for intracranial depth electrode mapping which requires brain surgery to place the depth electrodes to monitor for epileptic onset foci for consideration of future neuromodulation, resection, or ablation. This intracranial monitoring procedure is the platform for electrophysiological and neurochemical measurements and recordings we propose here. Importantly, we will only perform research recordings from sites that will necessarily be damaged by the clinical procedures, and due to the unknown epileptic foci, will later be deemed either healthy or epileptic tissue.

Cognitive processing occurs very rapidly over functionally organized networks that can be distributed among multiple brain areas. Consequently, understanding such complex functions requires the ability to map neuronal activity with high spatial and temporal resolution. Unfortunately, most noninvasive methodologies for recording neuronal activity have either high spatial or temporal resolution, but not both. However, electrocorticography (ECoG) offers the unique ability to record neuronal activity with both high spatial resolution (single-cell activity) and high temporal resolution (sub-millisecond time-scale).

Additionally, certain behaviors are uniquely human, including complex motor control, executive function, language processing, and speech generation. Many of these behaviors and their neural underpinnings are impossible to study in other species. If we are to improve treatments for human neurological and psychiatric conditions, it is critical to study them directly in humans. Patients already undergoing neurological surgery for functional brain mapping (Phase II epilepsy monitoring) offer the rare opportunity to test the neural underpinnings of these uniquely human behaviors via direct neurophysiological recordings. Moreover, ECoG and MER offer the ability to stimulate and record from multiple cortical and subcortical regions. Microstimulation allows for a more complete assessment of both the functional connectivity among isolated brain regions and the causal role(s) of these regions in cognition and behavior.

Similar work using intracranial recordings in humans has already enhanced our understanding of human cognition both in health and disease. For example, it has helped identify the neural correlates of human memory, language, error monitoring and behavioral adjustment and emotion. This work has helped to develop breakthroughs toward enhancing and restoring cognitive function in humans.

These studies do not put the patients at additional risk as the electrode placement is already required for the treatment of treatment resistant epilepsy.

There are several FDA approved electrodes for intracranial recording and monitoring. One available depth electrode used for clinical purposes is AdTech's "All-in-one Macro-Micro" electrode, where the micro contacts are radially spaced on the body of the depth electrode. Other electrodes, such as commercially available Behnke Fried electrode with clinical contacts and research microwires, are FDA approved for standard-of-care use side-by-side with clinical research recordings.

Currently, there is no technology available that will permit simultaneous sub-second measurements of dopamine, serotonin, and norepinephrine in the human brain; however, one of the collaborating scientists (Montague) has recently developed a novel approach that enables real-time measurements of dopamine and serotonin using carbon fiber micro-sensors and a machine learning based approach to fast scan cyclic voltammetry. Further, preliminary evidence from that investigators' lab suggests that this technology may be extended to simultaneously measure dopamine, serotonin, and norepinephrine in the human brain. The electrode and the algorithm (which uses as input the currents recorded by the electronic equipment connected to the electrode and is not necessary for the functioning of the electrode) are not medical devices and are used in this research for purely scientific reasons - not medical purposes.

Here, we propose to deploy a new recording protocol in combination with an FDA approved micro-sensor assembly that will enable simultaneous measurements dopamine, serotonin, and norepinephrine micro-fluctuations with sub-second temporal resolution in the human brain. If successful, the proposed work could provide a significant technological advance for neuroscience research in human brain function and behavior, with potential translational impact in areas including in neurosurgery, neurology, and psychiatry.

Background to electrochemical measurement approach. The critical measurement approach that enables simultaneous electrochemical detection of dopamine, serotonin, and norepinephrine is an electrochemical method called "fast scan cyclic voltammetry". This approach has been utilized in rodents and rodent brain tissue for over 25 years. Briefly, a voltage is applied to a carbon fiber microelectrode. If this voltage is greater than or equal to the oxidation potential of a chemical species, then an electrochemical oxidation reaction takes place and the transfer of electrons (to the carbon fiber) is measured as a change in current. By quickly scanning over a range of applied potentials (e.g., -0.6V to +1.4V and back to -0.6V at a scan rate of 400V/s), a range of electrochemical currents can be detected. We have developed a machine learning based algorithm that allows us to infer the chemical species' identity and concentration from this induced electrochemical spectrum. Prior reports demonstrate that we can continuously monitor dopamine, serotonin, and norepinephrine micro-fluctuations with 100ms temporal resolution, which is orders of magnitude faster and with direct chemical specificity better that existing non-invasive measurement modalities like fMRI and PET and invasive approaches like microdialysis. The algorithm is not intended for clinical or medical use and is strictly used as stated.

The clinical importance of investigating the action of the neurotransmitters dopamine, serotonin, and norepinephrine is perhaps best highlighted by the pharmaceuticals used to treat major psychiatric conditions like depression, anxiety disorders, chronic pain, attention deficit disorders, and nicotine addiction. Selective serotonin reuptake inhibitors (SSRIs) are used to treat depression and anxiety; Norepinephrine and Serotonin reuptake inhibitors (NSRIs) are used to treat depression and chronic pain; Norepinephrine and dopamine reuptake inhibitors are used to treat depression, attention deficit disorders, and have been used as an aid to smoking cessation; and Norepinephrine reuptake inhibitors (NRIs) have been used to treat depression, narcolepsy, attention deficit hyperactivity disorder, as an aid to weight loss, and anxiety disorders characterized by low arousal. Furthermore, abused substances (e.g., cocaine, nicotine, alcohol, and opiates) are known to alter the subtle balance between neurotransmitter release and reuptake in model organisms.

From a basic science perspective, the investigators believe that dopamine is critical for reward processing and motivated behavior, serotonin for processing aversive stimuli and mood regulation, and norepinephrine for regulating states of arousal and attention. These neurotransmitters are released from neurons located in the brain stem (serotonin and norepinephrine) and midbrain (dopamine) whose axon terminals distribute and broadcast these signals throughout the brain including targets throughout the cortex (dopamine, serotonin, and norepinephrine), basal ganglia (dopamine and serotonin), hippocampus (dopamine and serotonin), and amygdala (dopamine, serotonin, and norepinephrine). While it is clear that these systems are critical, most of what is known comes from model organism research at timescales too slow to understand how rapid, real-time fluctuations in these signals contribute healthy human cognition, decision-making, and behavior.

We also have a very limited understanding of how dopamine, serotonin, and norepinephrine systems interact. In any given brain region, it may be expected that there are one, two, or all three of these neurotransmitter systems contributing to the local neural information processing. In the human brain (and non-human primate brain) we know little about how the density of release sites or the dynamics of release change with psychiatric conditions or the medications used to treat them. This lack of knowledge does not stem from a lack of interest in the neuroscience, neurology, psychiatry, or neurosurgery disciplines; rather, the necessary technology and research paradigm has not been available. This proposal seeks to take the first steps in developing novel hardware (micro-sensor assembly) and pair it with the Dr Montague's machine learning based approach to fast scan cyclic voltammetry to simultaneously measure continuous sub-second micro-fluctuations of dopamine, serotonin, and norepinephrine in the human brain. (to study basic properties of these neuromodulator's dynamics in human subjects.)

Simultaneous sub-second measurements of dopamine, serotonin, and norepinephrine in the human brain would allow investigators to monitor how these three neurotransmitters fluctuate in real-time. Such technology could potentially some day be used to develop real-time biomarkers of dynamic brain activity in disease specific brain areas, which may be used diagnostically or prognostically in psychiatry (e.g., depression or OCD) and neurology (e.g., Parkinson's disease or epilepsy) and neurosurgery (e.g., deep brain stimulation electrode placement or lesion/tumor resection boundaries). Further, such measurements could be used to assess exactly how drugs (clinical treatments or abused substances) alter the function of these neuromodulatory systems in real-time in the human brain. Finally, such technology could provide a breakthrough in intracranial neuroscience research into the basic neural mechanisms underlying decision-making We also have a very limited understanding of how dopamine, serotonin, and norepinephrine systems interact. In any given brain region, it may be expected that there are one, two, or all three of these neurotransmitter systems contributing to the local neural information processing. In the human brain (and non-human primate brain) we know little about how the density of release sites or the dynamics of release change with psychiatric conditions or the medications used to treat them. This lack of knowledge does not stem from a lack of interest in the neuroscience, neurology, psychiatry, or neurosurgery disciplines; rather, the necessary technology and research paradigm has not been available. This proposal seeks to take the first steps in developing novel hardware (micro-sensor assembly) and pair it with the Dr Montague's machine learning based approach to fast scan cyclic voltammetry to simultaneously measure continuous sub-second micro-fluctuations of dopamine, serotonin, and norepinephrine in the human brain. (to study basic properties of these neuromodulator's dynamics in human subjects.)

Simultaneous sub-second measurements of dopamine, serotonin, and norepinephrine in the human brain would allow investigators to monitor how these three neurotransmitters fluctuate in real-time. Such technology could potentially some day be used to develop real-time biomarkers of dynamic brain activity in disease specific brain areas, which may be used diagnostically or prognostically in psychiatry (e.g., depression or OCD) and neurology (e.g., Parkinson's disease or epilepsy) and neurosurgery (e.g., deep brain stimulation electrode placement or lesion/tumor resection boundaries). Further, such measurements could be used to assess exactly how drugs (clinical treatments or abused substances) alter the function of these neuromodulatory systems in real-time in the human brain. Finally, such technology could provide a breakthrough in intracranial neuroscience research into the basic neural mechanisms underlying decision-making processes that may generally be affected in humans prone to poor health-related behaviors.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 80 years, inclusive.
* Patients who are candidates for electrode implantation due to pharmacologically intractable epilepsy, or other neurological/psychological disorders for which subdural electrode implantation may be clinically required for treatment.
* Patients competent to give informed consent/assent for the research protocol and parents of children under 18 who are competent to give informed consent on behalf of the child.
* Fluency in English (necessary for uniform cognitive testing).
* Committee approved candidates for brain surgery.
* Medications must be at stable doses for at least 1 month before surgery

Exclusion Criteria:

* Clinically significant cognitive dysfunction.
* Terminal illness associated with <12 month survival.
* Contraindication to MRI imaging, e.g., morbid obesity, metallic devices such as cardiac pacemakers, some aneurysm clips, or shrapnel.
* Current pregnancy or pregnancy planned during the course of the study.
* Cognitive function less than 2 standard deviations below normal on preoperative neuropsychological testing

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2022-09-07 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Neurotransmitter Concentration Fluctuation in Visual Memory | During Hospitalization - 1-2 weeks
  Neurotransmitter concentrations will be recorded through Fast Scan Cyclic Voltammetric methods during cognitive psychological tasks for visual memory administered on a laptop.
Neurotransmitter Concentration Fluctuation and Pupillary Diameter in Sustained Attention Tasks | During Hospitalization - 1-2 weeks
  Neurotransmitter concentrations will be recorded through Fast Scan Cyclic Voltammetric methods and and pupillary diameter will be observe with a pupillometer during cognitive psychological tasks for sustained attention administered on a laptop.
Neurotransmitter Concentration Fluctuation in Neuroeconomics Tasks | During Hospitalization - 1-2 weeks
  Neurotransmitter concentrations will be recorded through Fast Scan Cyclic Voltammetric methods during cognitive psychological tasks for neuroeconomics administered on a laptop.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Bina, MD, Principal Investigator — University of Arizona
Locations (1):
- Banner - University Medical Center, Phoenix campus, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be stored and collected on the University of Arizona REDCap and deidentified data will be shared with Arizona State University (ASU) and Virginia Tech (VT) researchers.
Supporting Information: Study Protocol
Time Frame: Data will be available for ASU and VT from initiation of the project, all the way through data analysis.
Access Criteria: Virginia Tech and ASU will have access to the de-identified data via encrypted email or the University of Arizona's REDCap EDM.